CLINICAL TRIAL: NCT01358396
Title: The Effect of Glycemic Control on Visual and Anatomical Outcomes in Response to Therapy for Diabetic Macular Edema.
Brief Title: Glycemic Control and Diabetic Macular Edema
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Tamer A Macky, Cario University
Other Study IDs: HB-DME-1
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2010-01

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema, Glycemic Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HBA1c
  Interventions: Other: Respond to therapy for diabetic macular edema

INTERVENTIONS:
Other: Respond to therapy for diabetic macular edema — Correlate HBA1c with visual acuity outcome to therapy.
  Other Names: Diabetic Macular Edema and Glycemic Control Using glycosylated hemoglobin

SUMMARY:
Does diabetic patients' glycemic control affect their response to laser and/or intravitreal injection therapy in terms of visual and anatomical outcomes.

DETAILED DESCRIPTION:
To evaluate the visual and anatomical response to therapy in patients with diabetic macular edema (DME) in relation to their glycemic control.

Patients with DME with central foveal thickness (CFT) > 250µm with no proliferative disease had their glycosolated hemoglobin (HbA1c) measured at baseline and 3 months. CFT by optical coherence tomography, and best corrected visual acuity (BCVA) in logMARs were measured at baseline, 1, and 3 months. Exclusion criteria: laser or intravitreal injections within 6 months, hard exudates within 500um of the foveal center, or macular traction. Therapy included laser and intravitreal anti VEGFs. HbA1c graded as: G1=<7%, G2= 7-7.9%, G3= 8-8.9%, G4 = >9%; and as: low <8%, high ≥ 8%.

ELIGIBILITY:
Inclusion Criteria:

* Central foveal thickness more than 250 microns

Exclusion Criteria:

* Proliferative Diabetic Retinopathy.
* Traction Macular Membranes
* Previous Laser or intravitreal injections within 6 months.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients with macular edema with central foveal thickness more than 250 microns and no proliferative changes.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Correlate baseline HBA1c to the visual outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt